CLINICAL TRIAL: NCT01279460
Title: Evaluation of Aortic Stiffness in CKD II to IV
Brief Title: Aortic Stiffness in Chronic Kidney Disease Stage 2 to 4
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Department of Nephrology, Klinikum rechts der Isar, München (Unknown)
Responsible Party: PD. Dr. med. Marcus Baumann, M.D., PhD, Technical University of Munich, Klinikum rechts der Isar, Department of nephrology
Other Study IDs: Munich-CKD-PWA
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Decline in Renal Function
Keywords: chronic kidney disease; CKD; pulse wave velocity; PWV
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CKD Cohort of patients with renal insufficiency: patients with renal insufficiency grade II-IV

SUMMARY:
This study aimed to investigate in a cohort with chronic kidney disease the longitudinal relationship between aortic stiffness and renal function and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* CKD 2-4

Exclusion Criteria:

* pregnancy
* history of malignant disease with a prognostic life expectancy less than 24 months
* missing of written and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were enrolled in a prospective study of vascular stiffness and CV risk in patients with CKD stages 2 to 4. They were predominantly recruited from outpatients attending nephrology clinics at the Klinikum rechts der Isar der Technischen Universität München and at a private nephrological clinic in Weissenburg October 2007 to December 2008.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
combined renal end-point (>25% decline in renal function or start of renal replacement therapy) | 24 months

SECONDARY OUTCOMES:
mortality | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Baumann, M.D. PhD, Principal Investigator — Klinikum rechts der Isar of the Technical University Munich
Locations (2):
- Germany (2):
  - Klinikum rechts der Isar, München, Bavaria
  - Klinikum Weissenburg, Weißenburg in Bayern, Bavaria

REFERENCES:
- [Background] Pan CR, Roos M, Schmaderer C, Lutz J, Wang JG, Heemann U, Baumann M. Interrelationship between aortic stiffness and proteinuria in chronic kidney disease. J Hum Hypertens. 2010 Sep;24(9):593-9. doi: 10.1038/jhh.2009.108. Epub 2010 Jan 28. PMID 20107490
- [Background] Townsend RR, Wimmer NJ, Chirinos JA, Parsa A, Weir M, Perumal K, Lash JP, Chen J, Steigerwalt SP, Flack J, Go AS, Rafey M, Rahman M, Sheridan A, Gadegbeku CA, Robinson NA, Joffe M. Aortic PWV in chronic kidney disease: a CRIC ancillary study. Am J Hypertens. 2010 Mar;23(3):282-9. doi: 10.1038/ajh.2009.240. Epub 2009 Dec 17. PMID 20019670